CLINICAL TRIAL: NCT01485484
Title: Development and Validation of a NIRS-based Sinusitis Screening
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Naveen Bhandarkar, M.D., Assistant Clinical Professor, Department Otolaryngology, University of California, Irvine
Other Study IDs: 20118295
Record Dates: First submitted 2011-10-28; First posted 2011-12-05 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Sinusitis
MeSH Terms: conditions — Sinusitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sinus: Optic imaging use near-infrared trans-illumination methods
  Interventions: Device: Optic imaging use near-infrared trans-illumination methods

INTERVENTIONS:
Device: Optic imaging use near-infrared trans-illumination methods — Optic imaging use near-infrared trans-illumination methods

SUMMARY:
The research at University of California Irvine, Beckman laser institute and Praxis Biosciences Incorporation, develope near-infrared trans-illumination methods. The optical imaging tool that can determine acute sinusitis and the response to treatment therapy.

DETAILED DESCRIPTION:
In the United States, approximately one in seven people develop sinusitis each year, and 20 million cases of acute bacterial sinusitis become chronic to require medical treatment. The optic light from the illumination wand travelled through the pallet into the sinuses and exited the face. The optic device can determine air-filled and fluid/tissue-filled spaces in the sinus cavity during clinical exam.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years of age and older
* Subject with normal sinus
* Subject who has been diagnosed and confirm by their physician

Exclusion Criteria:

* Younger than 18 years old
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be selected from outpatient clinic at Otolaryngology Clinic at the University of California, Irvine Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2011-07-28 (Actual); Primary Completion 2015-07-07 (Actual); Study Completion 2015-07-07 (Actual)

PRIMARY OUTCOMES:
Sinus Health | up to 4 weeks
  Assessment of sinusitis

CONTACTS AND LOCATIONS:
Overall Officials: Naveen Bhandarkar, MD, Principal Investigator — University of California, Irvine
Locations (1):
- UCI Beckman Laser Medical Clinic, Irvine, California, United States